CLINICAL TRIAL: NCT00775606
Title: A Phase 4 Study of the Effect on Immune Reconstitution of a Lopinavir/Ritonavir-Based Versus an Efavirenz-based HAART (Highly Active Antiretroviral Therapy) Regimen in Antiretroviral-Naïve Subjects With Advanced HIV Disease
Brief Title: Immune Reconstitution of Lopinavir/Ritonavir-Based vs Efavirenz-based HAART in Advanced HIV Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped 12/2010 due to poor enrollment. Only 15 of 60 needed enrolled.
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Chicago (Other); University of Illinois at Chicago (Other); Ruth M. Rothstein CORE Center (Other); Abbott (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Beverly E. Sha, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICE-001
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Acquired Immune Deficiency Syndrome
Keywords: AIDS, HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A/Lopinavir/ritonavir (Active Comparator): Subjects randomized to Arm A initiated Lopinavir 400 mg/ritonavir 100 mg BID + emtricitabine 200 mg/tenofovir 300 mg QD
  Interventions: Drug: Lopinavir 400 mg/ritonavir 100 mg
- ARM B/Efavirenz (Active Comparator): Subjects randomized to Arm B initiated Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg QD
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Lopinavir 400 mg/ritonavir 100 mg — Lopinavir 400 mg/ritonavir 100 mg fixed dose combination BID + emtricitabine 200 mg/tenofovir 300 mg fixed dose combination QD
  Other Names: Kaletra; Truvada
  Arms: ARM A/Lopinavir/ritonavir
Drug: Efavirenz — Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg fixed dose combination QD
  Other Names: Atripla
  Arms: ARM B/Efavirenz

SUMMARY:
The ideal anti-HIV medications for patients with advanced HIV disease is unknown. There is evidence that anti-HIV regimens that contain protease inhibitors can enhance immune function better than regimens that do not contain protease inhibitors. This is a study that will determine the difference in immune enhancement capabilities between an anti-HIV regimen that contains the protease inhibitor - lopinavir-ritonavir, and a regimen that contains efavirenz. Both medications are recommended as first line treatments for HIV-infected patients. This study will recruit HIV-positive patients that need to start anti-HIV treatment because their CD4+ T-cells are below 200. The usual threshold for starting treatment is a CD4+ T-cell less than 350. Subjects will be randomized to treatment with either an anti-HIV regimen that contains lopinavir-ritonavir or a regimen that contains efavirenz. The study will determine the difference in immune reconstitution over 24 weeks of treatment with study medications. Among the immune parameters that will be measured is the ability of each subject to respond to vaccination with the tetanus-diphtheria vaccine and the 23-valent pneumococcal vaccine. Both vaccines are also recommended for HIV-positive patients but HIV-positive patients tend to have a lower response rate to these vaccines.

DETAILED DESCRIPTION:
DESIGN: ICE-001 is a phase IV, randomized, two-arm unblinded study, comparing the effect on immune reconstitution of open-label ritonavir (RTV)-enhanced lopinavir (LPV) to efavirenz (EFV), in combination with daily emtricitabine (FTC)/tenofovir (TDF) as initial therapy for HIV-1 infection in HIV-infected treatment naïve subjects with CD4+ T-cells less than 200 cells/ml.

DURATION: Subjects will participate in ICE-001 for approximately 48 weeks after starting study treatment.

SAMPLE SIZE: ICE-001 will enroll 60 subjects (30 per treatment arm).

POPULATION: HIV-1-infected, antiretroviral (ARV) drug-naïve (≤7 days of ARV treatment at anytime prior to study entry) men and women between18 to 60 years of age with plasma HIV-1 RNA levels >1000 copies/mL and CD4+ T-cell counts < 200 cells/ml obtained within 90 days prior to study entry.

STRATIFICATION: Subjects will be stratified at screening based on plasma HIV-1 RNA levels <100,000 and ≥100,000 copies/mL.

REGIMEN: At entry subjects will be randomized to one of the following:

* ARM A: LPV 400 mg/RTV 100 mg BID + FTC 200 mg/TDF 300 mg QD
* ARM B: EFV 600 mg QD/FTC 200 mg/TDF 300 mg fixed dose combination QD

The objective is to determine the differences in the degree of immune reconstitution in HIV-infected patients with a CD4+ T-cell count < 200 cells/ml who initiated treatment with LPV/RTV + FTC/TDF compared to EFV/FTC/TDF.

Study visits will occur at screening, pre-entry, entry and weeks 1, 4, 8, 12, 24 and 48 after study entry. Study medications will be provided at entry after randomization. At most study visits, clinical assessments, including histories, physical exams and determination of drug adherence, will occur. Blood for hematologic and metabolic safety assessments and for the assessment of immune parameters will be obtained. Immune parameters that will be measured include levels of T-cell apoptosis, maturation and activation. Frequencies of various T-cell subsets and other lymphocyte populations will also be done. Response to vaccination with tetanus-diphtheria vaccine and 23-valent pneumococcal polysaccharide vaccine (both given at week 8) will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection
2. The absence of exclusionary resistance mutations on a genotypic resistance assay
3. Antiretroviral (ARV) drug-naïve
4. Screening HIV-1 RNA >1000 copies/mL
5. Screening CD4+ T-cell count < 200 cells/ml
6. Laboratory values obtained within 30 days prior to study entry.

   * Absolute neutrophil count (ANC) >500/mm3
   * Hemoglobin >8.0 g/dL
   * Platelet count >40,000/mm3
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase <5 x ULN
   * Total bilirubin <2.5 x ULN
   * Calculated creatinine clearance ≥60 mL/min (by Cockcroft-Gault equation)
7. For women of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to initiating study medications.
8. Contraception requirements
9. Men and women age >18 years and < 60 years.
10. Ability and willingness of subject or legal guardian/representative to give written informed consent.

Exclusion Criteria:

1. Currently breast-feeding.
2. Use of immunomodulators, vaccines, growth hormone, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.
3. Known allergy/sensitivity to study drugs, pneumococcal polysaccharide vaccine, tetanus-diphtheria vaccine
4. Receipt of pneumococcal polysaccharide vaccine or tetanus-diphtheria vaccine in the past 5 years.
5. Active drug or alcohol use or dependence
6. Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 14 days prior to study entry.
7. Requirement for any current medications that are prohibited with any study treatment.
8. Evidence of any major resistance-associated mutation on any genotype or evidence of significant resistance on any phenotype performed at any time prior to study entry
9. Current or anticipated imprisonment or involuntary incarceration in a medical facility for psychiatric or physical (e.g., infectious disease) illness
10. History of, or current bipolar disorder, major depression, schizophrenia or other psychotic disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan R. Tenorio, M.D., Study Chair — Rush University Medical Center
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois

REFERENCES:
- [Result] Pitrak DL, Novak RM, Estes R, Tschampa J, Abaya CD, Martinson J, Bradley K, Tenorio AR, Landay AL. Short communication: Apoptosis pathways in HIV-1-infected patients before and after highly active antiretroviral therapy: relevance to immune recovery. AIDS Res Hum Retroviruses. 2015 Feb;31(2):208-16. doi: 10.1089/aid.2014.0038. Epub 2014 Nov 11. PMID 25386736

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects withdrew participation prior to starting study
Groups:
- ARM A/Lopinavir-ritonavir: Subjects randomized to Arm a will initiate Lopinavir 400 mg/ritonavir 100 mg BID + emtricitabine 200 mg/tenofovir 300 mg QD
- ARM B/Efavirenz: Subjects randomized to Arm B will initiate Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg QD
Period: Overall Study
Arm/Group | ARM A/Lopinavir-ritonavir | ARM B/Efavirenz
Started | 8 | 5
Completed | 5 | 5
Not Completed | 3 | 0
Not completed — Study sponsor terminated funding | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARM A: Subjects randomized to Arm a will initiate Lopinavir 400 mg/ritonavir 100 mg BID + emtricitabine 200 mg/tenofovir 300 mg QD
- ARM B: Subjects randomized to Arm B will initiate Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg QD
- Total: Total of all reporting groups
Arm/Group | ARM A | ARM B | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.4) | 30.6 (7.1) | 33 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: CD4+ (Cluster of Differentiation 4) T-cell Apoptosis
Description: Change in the percentage of naive CD4 T-cells undergoing apoptosis as measured by propidium iodide staining. This is a lab test that measures the percentage of naive CD4 T-cells that are undergoing cell death. The change in this measure is obtained by determining the difference between the percentage of naive CD4 T-cells undergoing apoptosis at week 24 of treatment and the percentage undergoing apoptosis at baseline.
Time Frame: 24 weeks from treatment initiation (baseline and week 24)
Measure: Mean (Standard Deviation); unit: per cent
Arm/Group | ARM A/Lopinavir-ritonavir | ARM B/Efavirenz
Number analyzed (Participants) | 5 | 5
per cent | -12.33 (12.34) | -8.01 (7.97)

2. Secondary Outcome: CD4+ T-cell Change
Description: This measures the change in CD4+ T-cells from baseline to week 24 of treatment.
Time Frame: 24 weeks after treatment initiation (baseline and week 24)
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | ARM A/Lopinavir-ritonavir | ARM B/Efavirenz
Number analyzed (Participants) | 5 | 5
cells/mm3 | 176.83 (101.39) | 102.6 (150.45)

3. Secondary Outcome: Naive, Central Memory, Effector Memory, and T Reg CD4+ T-cell Frequency
Description: Naive, central memory, effector memory, and T reg CD4+ T-cell frequency at baseline
Time Frame: baseline measurements
Population: 11 subjects contributed to the baseline data (6 randomized to lopinavir/ritonavir and 5 randomized to efavirenz).
Measure: Mean (Full Range); unit: percentage of cells
Groups:
- ARM A Lopinavir/Ritonavir: Subjects randomized to Arm A initiated Lopinavir/ritonavir 400/100 mg po bid
- ARM B Efavirenz: Subjects randomized to Arm B initiated Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg QD.
Arm/Group | ARM A Lopinavir/Ritonavir | ARM B Efavirenz
Number analyzed (Participants) | 6 | 5
percentage of cells
  Mean percentage of naive CD4+ T cells at baseline | 32.67 [23.73 to 45.54] | 24.70 [1.66 to 38.54]
  Mean percentage of central memory CD4+ T cells at baseline | 11.54 [5.09 to 16.43] | 9.02 [6.03 to 11.49]
  Mean percentage of effector memory CD4+ T cells at baseline | 36.44 [24.86 to 46.3] | 47.32 [31.25 to 64.31]
  Mean percentage of CD4+ Treg cells at baseline | 7.35 [1.46 to 16.87] | 6.96 [3.57 to 12.78]

4. Secondary Outcome: Naive, Central Memory, Effector Memory, and T Reg CD4+ T-cell Frequency
Description: Naive, central memory and effector memory, and T reg CD4+ T-cell frequency at week 24
Time Frame: week 24 measurements
Population: 10 subjects contributed to the week 24 data (6 randomized to lopinavir/ritonavir and 4 randomized to efavirenz).
Measure: Mean (Full Range); unit: percentage of cells
Groups:
- ARM B Efavirenz: Subjects randomized to Arm B initiated Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg QD.
  5 subjects contributed to the baseline data but only 4 subjects contributed to the week 24 data.
Arm/Group | ARM A Lopinavir/Ritonavir | ARM B Efavirenz
Number analyzed (Participants) | 6 | 4
percentage of cells
  Mean percentage of naive CD4+ T cells at week 24 | 29.08 [17.8 to 47.25] | 25.73 [1.82 to 49.13]
  Mean percentage of central memory CD4+ T cells at week 24 | 10.89 [3.83 to 22.37] | 8.28 [5.48 to 11.03]
  Mean percentage of effector memory CD4+ T cells at week 24 | 34.98 [24.37 to 43.37] | 44.82 [21.55 to 69.53]
  Mean percentage of CD4+ Treg cells at week 24 | 5.58 [1.6 to 8.63] | 5.51 [4.7 to 6.52]

5. Secondary Outcome: Activation and Proliferation of CD4+ and CD8+ T-cell Frequencies
Description: Activation and proliferation of CD4+ and CD8+ T cells were measured at baseline
Time Frame: baseline measurements
Population: 11 subjects contributed to the baseline data (6 randomized to lopinavir/ritonavir and 5 randomized to efavirenz).
Measure: Mean (Full Range); unit: percentage of cells
Groups:
- ARM A Lopinavir-ritonavir: Subjects randomized to Arm A initiated Lopinavir 400 mg/ritonavir 100 mg BID + emtricitabine 200 mg/tenofovir 300 mg QD
Arm/Group | ARM A Lopinavir-ritonavir | ARM B Efavirenz
Number analyzed (Participants) | 6 | 5
percentage of cells
  Activation of CD4+ T cells at baseline | 12.85 [4.52 to 16.11] | 12.35 [5.61 to 16.92]
  Activation of CD8+ T cells at baseline | 34.61 [21.25 to 41.21] | 33.57 [11.36 to 59.10]
  Proliferation of CD4+ T cells at baseline | 1.21 [0.73 to 2.11] | 1.25 [0.56 to 2.20]
  Proliferation of CD8+ T cells at baseline | 1.39 [0.71 to 2.49] | 1.25 [0.58 to 2.41]

6. Secondary Outcome: Activated and Regulatory CD4+ and CD8+ T-cell Frequencies
Description: Activation of CD4+ and CD8+ T cells were measured at week 24
Time Frame: week 24 measurements
Population: 10 subjects contributed to the week 24 data (6 randomized to lopinavir/ritonavir and 4 randomized to efavirenz).
Measure: Mean (Full Range); unit: percentage of cells
Groups:
- ARM B Efavirenz: Subjects randomized to Arm B initiated Efavirenz 600 mg/emtricitabine 200 mg/tenofovir 300 mg QD
  5 subjects contributed to the baseline data but only 4 contributed to the week 24 data
Arm/Group | ARM A Lopinavir-ritonavir | ARM B Efavirenz
Number analyzed (Participants) | 6 | 4
percentage of cells
  Activation of CD4+ T cells at week 24 | 8.70 [3.42 to 12.39] | 7.39 [6.12 to 10.74]
  Activation of CD8+ T cells at week 24 | 20.92 [6.72 to 29.97] | 17.17 [6.08 to 24.24]
  Proliferation of CD4+ T cells at week 24 | 0.47 [0.25 to 0.68] | 0.52 [0.24 to 0.8]
  Proliferation of CD8+ T cells at week 24 | 0.81 [0.21 to 3.08] | 0.48 [0.16 to 0.97]

7. Secondary Outcome: Response to Immunization With Pneumococcus Polysaccharide and Tetanus-diphtheria Vaccines
Description: Response to immunization with pneumococcus polysaccharide and tetanus-diphtheria vaccines was not done due to small sample size
Time Frame: 4 weeks after treatment initiation
Population: Response to PPSV23 and Td vaccines was not performed due to the small sample size.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 24
Arm/Group | ARM A/Lopinavir-ritonavir | ARM B/Efavirenz
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 1/8 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A/Lopinavir-ritonavir (N=8) | ARM B/Efavirenz (N=5)
Grade 3 elevation in ALT (Hepatobiliary disorders) | 1 (1) | 0 (0) — Not related to study treatment. Related to alcohol use.

LIMITATIONS AND CAVEATS:
Study was terminated due to the slow recruitment and the small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No